CLINICAL TRIAL: NCT03819673
Title: A Computerised Decision-Support Tool for Health Professionals for the Prevention and Treatment of Childhood Obesity
Brief Title: Computerised Decision-Support Tool for Childhood Obesity Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, Yannis Manios, Principal Investigator, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: e-tool for childhood obesity
Record Dates: First submitted 2019-01-25; First posted 2019-01-28 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Childhood Obesity
Keywords: Personalised; Nutrition; Intervention; Children; Obesity; Health professionals
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (IG) (Experimental): Care based on the computerised decision-support tool
  Interventions: Behavioral: Intervention Group Care
- Control Group (CG) (No Intervention): Usual care advice by primary care provider or dietitian of participating hospital

INTERVENTIONS:
Behavioral: Intervention Group Care — children's assessment, setting weight management goals, provision of personalised meal plans, personalised diet and lifestyle optimization advice recommendations to children and their families, periodic re-evaluation every 3 or 6 months
  Arms: Intervention Group (IG)

SUMMARY:
The objective of the present study was to examine the effectiveness of a computerised decision-support tool, developed to assist paediatric clinicians in delivering personalised nutrition and lifestyle optimization advice to children and their families, as a means of childhood obesity management.

DETAILED DESCRIPTION:
The objective of the present study was to examine the effectiveness of a computerised decision-support tool, developed to assist paediatric clinicians in delivering personalised nutrition and lifestyle optimization advice to children and their families, as a means of childhood obesity management.

The effectiveness of the decision support tool was assessed through a pilot randomized controlled intervention trial (RCT). The RCT was initiated on May 2018 and was conducted in the Endocrinology Department of the "P. A. Kyriakou" Children's Hospital and in the Division of Endocrinology, Metabolism, and Diabetes of the "Aghia Sophia" Children's Hospital in Athens, Greece.

Sixty-five overweight or obese children that were eligible to participate in the RCT, were randomly and equally allocated to two study groups. Those children that were randomly allocated to the intervention group (IG), were examined by health professionals (i.e. paediatricians, paediatric endocrinologists and a dietitian) who were trained in the use of the decision support tool. The latter assisted the medical professionals to assess children's weight status, to set appropriate weight management goals and provide personalised meal plans and/or recommendations to children and their families. On the contrary, those children that were randomly allocated to the control group (CG) received the usual care advice that is routinely provided to children in the two hospitals and includes child visits and follow-up appointments for weight checks with their primary care provider or dietitian.

The effectiveness of the intervention was evaluated through the collection of data at baseline and at a follow-up examination after 3 months.

All data were uploaded to the decision-support tool, which analysed them and extracted a report with the child's assessment, as well as with personalised diet and lifestyle optimization recommendations. More specifically, the decision support tool proposed personalised weekly meal plans adjusted to the estimated energy requirements calculated for each child, as well as personalised diet and lifestyle optimization advice recommendations for the child and/or the entire family. Lastly, the decision support tool suggested a periodic re-evaluation every 3 or 6 months depending on the child's current weight status, the presence of obesity-related comorbidity in children and the presence of obesity in at least one or both parents.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-12 years old
* Overweight status or obesity (i.e. BMI-for-age > 85th percentile)

Exclusion Criteria:

* Age range not within the inclusion criteria

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yannis Manios, Professor, Principal Investigator — Harokopio University, Athens, Greece; George Moschonis, Associate Professor, Principal Investigator — La Trobe University, Bundoora, VIC 3086, Australia
Locations (1):
- Harokopio University of Athens, Kallithea, Attica, Greece